CLINICAL TRIAL: NCT06742086
Title: A Bioavailability and Food Effect Study of Venetoclax New Tablet Formulation 2.0 in Healthy Female Subjects
Brief Title: A Study to Evaluate the Bioavailability and Food Effects of Oral Venetoclax New Tablet Formulation 2.0 in Healthy Adult Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-277
Record Dates: First submitted 2024-12-17; First posted 2024-12-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Venetoclax; ABT-199; Venclexta; Venclyxto
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Stage 1: Sequence 1: Venetoclax (Experimental): Participants will receive commercial venetoclax following a high-fat meal (Regimen A), followed by venetoclax hot melt extrusion-03 (HME-03) dose A following a high-fat meal (Regimen B), followed by venetoclax HME-03 dose B following a high-fat meal (Regimen C), finally followed by venetoclax HME-03 dose A following fasting (Regimen D), as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax
- Stage 1: Sequence 2: Venetoclax (Experimental): Participants will receive Regimen B, followed by Regimen C, followed by Regimen A, finally followed by Regimen D, as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax
- Stage 1: Sequence 3: Venetoclax (Experimental): Participants will receive Regimen C, followed by Regimen A, followed by Regimen B, finally followed by Regimen D, as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax
- Stage 2: Sequence 1: Venetoclax (Experimental): Participants will receive Regimen A, followed by Regimen B, finally followed by Regimen C, as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax
- Stage 2: Sequence 2: Venetoclax (Experimental): Participants will receive Regimen B, followed by Regimen C, finally followed by Regimen A, as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax
- Stage 2: Sequence 3: Venetoclax (Experimental): Participants will receive Regimen C, followed by Regimen A, finally followed by Regimen B, as part of the approximately 18 month study duration.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Oral Tablet
  Other Names: ABT-199; Venclexta; Venclyxto

SUMMARY:
The objective of this study is to assess the bioavailability (BA) of venetoclax new high drug load hot melt extrusion-03 (HME-03) tablet formulation at two different tablet strengths relative to the commercial venetoclax tablet formulation under high-fat conditions in healthy female volunteers. Additionally, this study will assess the potential food effect on the BA of the venetoclax HME-03 tablet at the highest dosage strength.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) is 18.0 to 32.0 kg/m^2.
* Must either be: postmenopausal, permanently surgically sterile, or perimenopausal or premenopausal and practicing a method of birth control until at least 30 days after the last dose of study drug.
* Have CD19+ B-cell count > 150 cells/μL at screening.

Exclusion Criteria:

* History: of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, pulmonary, or hepatic diseases within the past 6 months that in the option of the investigator would adversely affect her participating in this study.
* History of any clinically significant sensitivity or allergy to any medication or food.
* History of or active medical condition(s) or surgical procedure(s) that might affect gastrointestinal motility, pH, or absorption [e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome, gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), cholecystectomy, vagotomy, bowel resection, etc.].

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 18 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Plasma Concentration (Cmax) of Venetoclax Hot Melt Extrusion-03 (HME-03) | Up to Approximately 18 Months
  Cmax of venetoclax HME-03.
Time to Cmax (Tmax) of Venetoclax HME-03 | Up to Approximately 18 Months
  Tmax of venetoclax HME-03.
Apparent Terminal Phase Elimination Constant (β) of Venetoclax HME-03 | Up to Approximately 18 Months
  β of venetoclax HME-03.
Terminal Phase Elimination Half-Life (t1/2) of Venetoclax HME-03 | Up to Approximately 18 Months
  t1/2 of venetoclax HME-03.
Area Under the Plasma Concentration-Time Curve from Time 0 Until the Last Measurable Concentration (AUCt) of Venetoclax HME-03 | Up to Approximately 18 Months
  AUCt of venetoclax HME-03.
Area Under the Plasma Concentration-Time Curve from Time 0 Until Infinity (AUCinf) of Venetoclax HME-03 | Up to Approximately 18 Months
  AUCinf of venetoclax HME-03.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Acpru /Id# 272979, Grayslake, Illinois
  - PPD Phase I Clinic /ID# 275754, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-277